CLINICAL TRIAL: NCT07219004
Title: A Prospective Multi-ceter Clinical Trail. Evaluating the Efficacy of Tri-layer Amnion/Chorion/Amnion (Artacent-AC) and Standard of Care in the Treatment of Chronic Lower Extremity Diabetic Ulcers.
Brief Title: Artacent Amniotic Tissue for Treatment of Chronic Lower Extremity Diabetic Ulcers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tides Medical (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POC-AC
Record Dates: First submitted 2025-10-15; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Lower Extremity Chronic Ulcers in Diabetics; Diabetic Foot Ulcer (DFU)
Keywords: Diabetic Foot Ulcers; Chronic foot ulcers; Plantar Ulcers; Lower Extremity Ulcers; Amniotic Tissues; HCT/P; 361 products; Q4190
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Leg Ulcer | interventions — Biological Dressings; cancer procoagulant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artacent-AC (Experimental): Artacent AC®is a HCT/P regulated solely as a "361 Product" and meets all criteria in 21 CFR 1271.10(a). The amnion and chorion layers are harvested from human placenta obtained during planned Caesarean sections. Tides Medical uses a proprietary process to clean the amniotic and chorion membranes. A Tri-Layered Amniotic Membrane (TLAM) is then formed by adding two outer layers of amnion with the stromal sides facing outward, separated by a middle chorion layer. TLAM is dried and cut into various sizes, packaged, and terminally sterilized.
  Artacent AC, like all other placental-derived products, is FDA cleared for homologous use through the 361 pathway. It is indicated for non-healing ulcers applied to a debrided, clean and uninfected ulcers as a wound cover.
  Interventions: Other: amniotic membrane

INTERVENTIONS:
Other: amniotic membrane — The intervention is a trial-layer human amnion/chorion/amnion composite graft
  Other Names: Chorion; Q4190; Amnion

SUMMARY:
This is study is to determine if A tri-layered dehydrated human amnion/chorion/amnion composite graft would help non-healing lower extremity diabetic ulcers to heal over a 12 week time period.

DETAILED DESCRIPTION:
This is study is to determine if A tri-layered dehydrated human amnion/chorion/amnion composite graft would help non-healing lower extremity diabetic ulcers to heal over a 12 week time period. During this trial the patient will undergo a screening period where SOC is used to see if the patient will respond and heal > 20% of the surface area in 2 weeks. if the patient can not heal more than 20% in two week the patient then will receive a trial-layered human amnion/chorion/amnion composite graft weekly for 12 week and precent wound area reduction and complete wound healing will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible to participate in the study if all the following conditions exist:

Potential subjects are required to meet all the following criteria for enrollment into the study.

1. Subjects must be at least 18 years of age or older,
2. Subjects must have a diagnosis of type 1 or 2 Diabetes mellitus.
3. At entry subjects must have a target ulcer with a minimum surface area of 0.7 cm2 and a maximum surface area of 20.0 cm2 measured post debridement with the MolecuLight Imaging HCT/P 361 .
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be full thickness without exposed bone.
7. The affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

   1. ABI between 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic.
8. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The subject must consent to using the prescribed off-loading method for the duration of the study.
11. The subject must agree to attend the weekly study visits required by the protocol.
12. The subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

* Subjects will be excluded from participation in the study if any of the following conditions exist:

  1. A subject known to have a life expectancy of < 6 months is excluded.
  2. The subject is excluded if the target ulcer is not secondary to diabetes.
  3. If the target ulcer is infected or if there is cellulitis in the surrounding skin, the subject is excluded.
  4. If there is evidence of osteomyelitis complicating the target ulcer, the subject is excluded.
  5. A potential subject cannot have an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
  6. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy is excluded.
  7. The topical application of steroids to the ulcer surface within one month of initial screening is not permitted.
  8. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
  9. If a subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit he/she is excluded.
  10. The subject is excluded if the surface area measurement of the Target ulcer decreases by 20% or more during the 2-week screening phase: the 2 weeks from the initial screening visit (S1) to the TV-1 visit during which time the subject received SOC.
  11. A Subject with an acute Charcot foot, or an inactive Charcot foot, that impedes proper offloading of the target ulcer is excluded.
  12. Women who are pregnant or considering becoming pregnant within the next 6 months are excluded.
  13. A potential subject with end stage renal disease requiring dialysis is excluded.
  14. A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days is excluded.
  15. A subject who in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments is excluded.
  16. A Subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Rate of wound closure by percent of complete epithelialization | 12 weeks
  complete wound closure measured by 100% epithelialization

SECONDARY OUTCOMES:
Percent area reduction | 12 weeks
  Precent of the wound which has been re-epithelialized

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, Principal Investigator — Serena Group
Locations (5):
- United States (5):
  - Three Rivers Wound and Hyperbaric Center, North Port, Florida
  - Serena Group Reseach Center, Buffalo, New York
  - Serena Group, Monroeville, Pennsylvania
  - The Serena Group Austin Research Center, Austin, Texas
  - El Campo Memorial Advanced Wound Care Clinic, El Campo, Texas

IPD SHARING:
Plan to Share IPD: No
Propritary study design